CLINICAL TRIAL: NCT02162771
Title: A Phase 3, Randomised, Parallel-Group, Active-Controlled, Double-Blind Study to Demonstrate Equivalence of Pharmacokinetics and Noninferiority of Efficacy for CT-P10 in Comparison With Rituxan, Each Administered in Combination With Cyclophosphamide, Vincristine, and Prednisone (CVP) in Patients With Advanced Follicular Lymphoma
Brief Title: To Demonstrate Equivalence of Pharmacokinetics and Noninferiority of Efficacy for CT-P10 in Comparison With Rituxan
Acronym: rituximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P10 3.3; 2013-004493-96 (EudraCT Number)
Record Dates: First submitted 2014-05-29; First posted 2014-06-13 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma, Follicular
Keywords: Advanced Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; CT-P10; Cyclophosphamide; Vincristine; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- CT-P10 (Experimental): Patient treated with CT-P10 (375 mg/m2 IV) in combination with cyclophosphamide (750 mg/m2 IV), vincristine (1.4 mg/m2 [max 2 mg] IV), and prednisone 40 mg/m2 orally) up to 8 cycles every 3 weeks during the Core Study Period.
  Patients having responses during Core Study Period treated with CT-P10 (375 mg/m2 IV) monotherapy up to 12 cycles every 2 months during the Maintenance Study Period.
  Interventions: Biological: CT-P10; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone
- Rituxan (Active Comparator): Patient treated with Rituxan (375 mg/m2 IV) in combination with cyclophosphamide (750 mg/m2 IV), vincristine (1.4 mg/m2 [max 2 mg] IV), and prednisone 40 mg/m2 orally) up to 8 cycles every 3 weeks during the Core Study Period.
  Patients having responses during Core Study Period treated with Rituxan (375 mg/m2 IV) monotherapy up to 12 cycles every 2 months during the Maintenance Study Period.
  Interventions: Biological: Rituxan; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Biological: Rituxan
  Other Names: Rituximab
  Arms: Rituxan
Biological: CT-P10
  Other Names: Rituximab
  Arms: CT-P10
Drug: Cyclophosphamide
Drug: Vincristine
Drug: Prednisone
  Other Names: Prednisolone

SUMMARY:
This study is a Phase 3 prospective, randomised, parallel-group, active controlled, double blind, multicentre, international study with 2 coprimary endpoints designed to demonstrate equivalence in pharmacokinetics (Part 1), as well as noninferiority in efficacy (Part 2), of CT-P10 to Rituxan when coadministered with CVP and to assess efficacy and safety in patients with advanced (stage III-IV) FL. Part 1 and Part 2 of the study will run in parallel.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female older than 18 years.
2. Patient has histologically confirmed FL according to the World Health Organization 2008 classification (Jaffe 2009); grades 1 to 3a based on local laboratory review.
3. Patient has at least 1 measurable tumour mass that has not previously been irradiated, and the mass must be:

   * greater than 1.5 cm in the longest dimension or
   * between 1.1 and 1.5 cm in the longest dimension and greater than 1.0 cm in the shortest axis
4. Patient has confirmed CD20+ lymphoma, as assessed by local laboratory review. (Tissue obtained within 6 months before Day 1 of Cycle 1 will be reviewed by a central independent reviewer to detect pathological type.)
5. Patient has Ann Arbor stage III or IV disease.

Exclusion Criteria:

1. Patient has received rituximab (or a rituximab biosimilar), cyclophosphamide, or vincristine.
2. Patient has allergies or hypersensitivity to murine, chimeric, human or humanised proteins, cyclophosphamide, vincristine, or prednisone.
3. Patient has evidence of histological transformation to high-grade or diffuse large B-cell lymphoma.
4. Patient has known central nervous system involvement.
5. Patient has received previous treatment for NHL:

   * Previous treatment including chemotherapy, radiotherapy, immunotherapy, and/or surgery (except previous biopsy)
   * All doses of corticoid therapy for treatment of NHL
   * Corticoid therapy during the previous 4 weeks from Day 1 of Cycle 1 with prednisone >20 mg per day for the treatment for any purpose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2016-01-12 (Actual); Study Completion 2018-12-29 (Actual)

REFERENCES:
- [Result] Kim WS, Buske C, Ogura M, Jurczak W, Sancho JM, Zhavrid E, Kim JS, Hernandez-Rivas JA, Prokharau A, Vasilica M, Nagarkar R, Osmanov D, Kwak LW, Lee SJ, Lee SY, Bae YJ, Coiffier B. Efficacy, pharmacokinetics, and safety of the biosimilar CT-P10 compared with rituximab in patients with previously untreated advanced-stage follicular lymphoma: a randomised, double-blind, parallel-group, non-inferiority phase 3 trial. Lancet Haematol. 2017 Aug;4(8):e362-e373. doi: 10.1016/S2352-3026(17)30120-5. Epub 2017 Jul 14. PMID 28712940
- [Derived] Buske C, Jurczak W, Sancho JM, Zhavrid E, Kim JS, Hernandez-Rivas JA, Prokharau A, Vasilica M, Nagarkar R, Kwak L, Kim WS, Lee S, Kim S, Ahn K, Ogura M. Long-term efficacy and safety of CT-P10 or rituximab in untreated advanced follicular lymphoma: a randomized phase 3 study. Blood Adv. 2021 Sep 14;5(17):3354-3361. doi: 10.1182/bloodadvances.2021004484. PMID 34477816
- See also: Related Info — http://www.celltrion.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 184 participants were screened for the study. Of those, 44 participants failed screening and 140 participants were enrolled in the study.
Period: Core Study Period (Part 2)
Arm/Group | CT-P10 | Rituxan
Started | 70 | 70
Completed | 62 | 62
Not Completed | 8 | 8
Not completed — Progressive Disease | 2 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Death | 1 | 0
Period: Maintenance Study Period (Part 2)
Arm/Group | CT-P10 | Rituxan
Started | 62 | 60 (Two subjects did not enter this period due to Withdrawal by subject and Non-responder, 1 for each.)
Completed | 46 | 38
Not Completed | 16 | 22
Not completed — Progressive Disease | 11 | 13
Not completed — Adverse Event | 3 | 3
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Stable Disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients (ITT population)
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P10 | Rituxan | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Median (Full Range); unit: years] | 57.0 [30 to 85] | 58.5 [26 to 84] | 57.5 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve at Steady State (AUCtau)
Description: AUCtau: Area under the plasma drug concentration-time curve within a dosing interval at steady state.
  PK sampling was done at pre-dose and 1 hour after the end of infusion (EOI) at Core Cycles 1-3 and 5-8. At Core Cycle 4 (i.e. steady state), intensive PK samplings were done as follows: predose, EOI, 1 hour after EOI, 24 hour after EOI, 168 hour after EOI, 336 hour after EOI, 504 hour after EOI. Lastly, one sample at any time of the end of treatment (EOT) 1 visit was obtained.
Time Frame: Core Cycle 4 (Week 12)
Population: Pharmacokinetic Population consisted of all patients who had at least 1 posttreatment PK concentration result after receiving at least 1 dose of study drug (CT-P10 or Rituxan) in Part 1. Patients considered outliers identified by a robust regression model (95% CI) were excluded from the analysis.
Measure: Geometric Mean (Standard Error); unit: h*ug/mL
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 50 | 56
h*ug/mL | 41002.43 (1.136) | 40099.08 (1.143)
Statistical Analysis 1: Comparison: CT-P10 vs Rituxan; Equivalence in AUCtau between CT-P10 and Rituxan; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed values were used to assess the bioequivalence between CT-P10 and Rituxan (bioequivalence range of 80% to 125%); ANCOVA; Country, gender, race, the value of ECOG status and the FLIPI score (0 to 2 versus 3 to 5) at baseline were fitted as covariates; Ratio of geometric least square means = 102.25, 90% CI 2-sided [94.05 to 111.17]

2. Primary Outcome: Maximum Serum Concentration at Steady State (Cmax,ss)
Description: Cmax,ss: Maximum concentration of drug in plasma at steady state on administering a fixed dose at equal dosing intervals.
  PK sampling was done at pre-dose and 1 hour after the end of infusion (EOI) at Core Cycles 1-3 and 5-8. At Core Cycle 4 (i.e. steady state), intensive PK samplings were done as follows: predose, EOI, 1 hour after EOI, 24 hour after EOI, 168 hour after EOI, 336 hour after EOI, 504 hour after EOI. Lastly, one sample at any time of the end of treatment (EOT) 1 visit was obtained.
Time Frame: Core Cycle 4 (Week 12)
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: ug/mL
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 53 | 56
ug/mL | 256.19 (1.115) | 254.49 (1.120)
Statistical Analysis 1: Comparison: CT-P10 vs Rituxan; Equivalence in Cmax,ss between CT-P10 and Rituxan; Test type: Equivalence — The 90% CIs of the ratios of geometric means of log-transformed transformed values were used to assess the bioequivalence between CT-P10 and Rituxan (bioequivalence range of 80% to 125%); ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric least square means = 100.67, 90% CI 2-sided [93.84 to 108.00]

3. Primary Outcome: Overall Response Rate (ORR) According to the 1999 International Working Group (IWG) Criteria
Description: ORR was defined as the proportion of patients with the best response of complete response (CR), unconfirmed complete response (CRu), or partial response (PR) by central review.
  Per 1999 IWG criteria, the disease status was assessed by using contrasted CT, and CR, CRu, and PR were defined as followings; CR=Disappearance of all clinical/radiographic evidence of disease: regression of lymph nodes to normal size, absence of B-symptoms, bone marrow involvement, and organomegaly, and normal LDH level; CRu=Regression of measurable disease: >=75% decrease in SPD of target lesions and in each target lesions. no increase in the size of non-target lesions, neither new lesion nor organomegaly measured; PR=Regression of measurable disease: >=50% decrease in SPD of target lesions and no evidence of disease progression.
Time Frame: During the Core Study Period (up to 8 cycles; Week 24)
Population: Efficacy population consisted of all patients who had at least 1 response evaluation after receiving at least 1 treatment cycle in the Core Study Period without any major protocol deviation that was relevant to the efficacy endpoint in Part 2.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 66 | 68
Participants | 64 | 63
Statistical Analysis 1: Comparison: CT-P10 vs Rituxan; Test type: Non-Inferiority — Non-inferiority margin of -7% was predefined; Point estimate difference = 4.3

4. Secondary Outcome: B-cell Kinetics (B-cell Depletion and Recovery)
Description: B-cell kinetics were demonstrated by median values of B-cell counts (Lower limit of quantification was 20 cells/uL).
Time Frame: Cycles 1 to 8 during the Core Study Period
Population: Pharmacodynamic (PD) population consisted of all patients who had at least 1 posttreatment PD result after receiving at least 1 dose of study drug (CT-P10 or Rituxan) without any major protocol deviation that was relevant to the PD endpoint in Part 2.
Measure: Median (Full Range); unit: cells/uL
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 70 | 70
cells/uL
  Core Cycle 1 (Predose): number analyzed (Participants) | 56 | 57
  Core Cycle 1 (Predose) | 92.5 [20 to 2890] | 62.0 [20 to 2890]
  Core Cycle 1 (1 hour after the end of infusion): number analyzed (Participants) | 44 | 55
  Core Cycle 1 (1 hour after the end of infusion) | 20.0 [20 to 1108] | 20.0 [20 to 51]
  Core Cycle 2 (Predose): number analyzed (Participants) | 60 | 60
  Core Cycle 2 (Predose) | 20.0 [20 to 1750] | 20.0 [20 to 2890]
  Core Cycle 3 (Predose): number analyzed (Participants) | 63 | 62
  Core Cycle 3 (Predose) | 20.0 [20 to 231] | 20.0 [20 to 35]
  Core Cycle 4 (Predose): number analyzed (Participants) | 59 | 61
  Core Cycle 4 (Predose) | 20.0 [20 to 51] | 20.0 [20 to 20]
  Core Cycle 5 (Predose): number analyzed (Participants) | 60 | 57
  Core Cycle 5 (Predose) | 20.0 [20 to 20] | 20.0 [20 to 20]
  Core Cycle 6 (Predose): number analyzed (Participants) | 60 | 61
  Core Cycle 6 (Predose) | 20.0 [20 to 33] | 20.0 [20 to 20]
  Core Cycle 7 (Predose): number analyzed (Participants) | 60 | 63
  Core Cycle 7 (Predose) | 20.0 [20 to 24] | 20.0 [20 to 20]
  Core Cycle 8 (Predose): number analyzed (Participants) | 61 | 59
  Core Cycle 8 (Predose) | 20.0 [20 to 20] | 20.0 [20 to 20]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious adverse events (SAEs) were to be collected from the date the ICF was signed until up to 30 days from last dose of the study drug, regardless of relationship to the study drug (a median follow up of 39.9 months).
Description: All TESAEs and non-serious AEs reported for more than 5% of the patients in either treatment group were summarized for the safety population. Safety population consisted of all patients who received at least 1 dose of the study drug (CT-P10 or Rituxan). Grading for severity and terminology of AEs were described according to the CTCAE Version 4.0.
Arm/Group | CT-P10 | Rituxan
Serious Adverse Events (participants affected / at risk) | 24/70 | 13/70
Other Adverse Events (participants affected / at risk) | 58/70 | 57/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P10 (N=70) | Rituxan (N=70)
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 4 | 1
Sialodenitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P10 (N=70) | Rituxan (N=70)
Hypertension (Vascular disorders) | 6 | 3
Fracture (Injury, poisoning and procedural complications) | 4 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 16 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 27 | 20
Dizziness (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 4 | 6
Hypoaesthesia (Nervous system disorders) | 6 | 2
Neuropathy peripheral (Nervous system disorders) | 10 | 12
Paraesthesia (Nervous system disorders) | 3 | 8
Asthenia (General disorders) | 5 | 8
Fatigue (General disorders) | 6 | 8
Oedema (General disorders) | 5 | 3
Pyrexia (General disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Constipation (Gastrointestinal disorders) | 12 | 10
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 9 | 7
Stomatitis (Gastrointestinal disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5
Fungal infection (Infections and infestations) | 4 | 4
Influenza (Infections and infestations) | 2 | 4
Lower respiratory tract infection (Infections and infestations) | 7 | 1
Sinusitis (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 18
Urinary tract infection (Infections and infestations) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality and non-disclosure agreement (CDA) was executed between Celltrion, Inc. and some PIs who have participated in publications funded by the sponsor for academic purposes for a period that is more than 180 days from the time submitted to the sponsor for review.